CLINICAL TRIAL: NCT07091409
Title: Neurobehavioral Mechanisms of Moral Reasoning: an EEG Study in Patients With Borderline Personality Disorder
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: BDP-MoDe
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-10

CONDITIONS: Borderline Personality Disorder (BPD)
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with BPD
- Healthy individuals

SUMMARY:
We will investigate social cognition in patients with Borderline personality disorder (BPD) combined with electroencephalographic (EEG) measures.

DETAILED DESCRIPTION:
We will investigate whether patients with Borderline personality disorder (BPD) show a negativity bias in evaluating social situations.

We will also asses emotional arousal, theory of mind (ToM) abilities, and inhibitory control in patients with BPD.

In addition to behavioral outcome variables, electroencephalographic (EEG) measures will be recorded. Healthy controls server as a control group.

ELIGIBILITY:
Inclusion Criteria:

BPD diagnosis BMI between 17.5 and 30 acute major depressive episode, psychotic symptoms, substance addiction or acute suicidal behavior

Exclusion Criteria:

neurological, metabolic, endocrine, autoimmune and CNS diseases, any other severe somatic diseases, and pregnancy or breastfeeding during the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BPD diagnosis and healthy participants
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Number of accidental harm scenarios misclassified as intentional | 20 Minutes
  Accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Psychiatry, CBF, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided